CLINICAL TRIAL: NCT02289066
Title: Impact of Periodontal Disease on Outcomes in Diabetes
Status: Completed | Type: Observational
Sponsor: University of Nevada, Reno (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1U54GM104944 (NIH); 1U54GM104944 (NIH)
Record Dates: First submitted 2014-10-23; First posted 2014-11-13 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Periodontal Disease; Diabetes Mellitus
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study examines how periodontal disease affects the complications of diabetes and how treatment for periodontal disease affects biomarkers associated with the complications of diabetes.

DETAILED DESCRIPTION:
The goal is to look for predictive factors of poor oral health and the impact of poor oral health on the complications of diabetes. The prevalence of periodontal disease among patients with diabetes is higher than in the general population. Periodontal disease is associated with dental loss and increased systemic inflammation which is associated with cardiovascular and bone disease. However, current evidence that treatment of POD will result in improvement of outcomes in patients with diabetes is mixed. Identifying patterns of disease and following biomarkers in patients with diabetes and periodontal disease will answer some of the questions and result in more appropriate recommendations and interventions with reduction in morbidity, mortality and healthcare cost.

This study will be conducted using a cross-sectional design. Investigators will survey 200 consecutive patients with diabetes during routine clinic visits using a questionnaire. Investigators will collect data on demographic information, socio-economic status, oral health status/care, diabetes history (duration, control and complications) and bone health. A subgroup of 24 participants with survey responses suggestive of periodontal disease will be selected to receive treatment for periodontal disease. We will measure their hemoglobin A1c and biomarkers before and after treatment and will compare their levels for changes with treatment. Investigators will analyze collected data using test of proportions, Student's t-test and multivariate regression analyses.

ELIGIBILITY:
Inclusion Criteria:

All patients 18 years or older with diabetes for more than 2 years who present for their regular clinic visit will be eligible for inclusion in the survey part of the study. Further criteria for enrollment into the subgroup (n = 24) will include; Inclusion criteria

* Answers on the questionnaire suggesting POD or gingivitis.
* At least 16 teeth in place
* On a stable treatment for their diabetes
* Hemoglobin A1c between 6 and 10

Exclusion Criteria:

* Treatment with anti-inflammatory medications
* Cigarette smoking
* Treatment with thiazolidinediones
* Previous diagnosis of osteoporosis or treatment for osteoporosis with FDA approved agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University of Nevada School of Medicine (Las Vegas) Internal medicine and endocrinology clinics
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in hemoglobin A1c | At enrollment, 3 months after enrollment and 6 months after enrollment.
biomarkers of inflammation (high sensitivity C - reactive protein and tumor necrosis factor - alpha) | At enrollment, 3 months after enrollment and 6 months after enrollment.
markers of bone turnover (bone specific alkaline phosphatase and C terminal | At enrollment, 3 months after enrollment and 6 months after enrollment.

SECONDARY OUTCOMES:
Evaluation of the relationship between periodontal disease and diabetes control and complications | At enrollment only

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Izuora, MD, MBA, Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada School of Medicine, Las Vegas, Nevada, United States

REFERENCES:
- [Background] 1. Centers for Disease Control and Prevention. National diabetes fact sheet: national estimates and general information on diabetes and prediabetes in the United States, 2011. Atlanta, GA: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, 2011.
- [Background] Boyle JP, Thompson TJ, Gregg EW, Barker LE, Williamson DF. Projection of the year 2050 burden of diabetes in the US adult population: dynamic modeling of incidence, mortality, and prediabetes prevalence. Popul Health Metr. 2010 Oct 22;8:29. doi: 10.1186/1478-7954-8-29. PMID 20969750